CLINICAL TRIAL: NCT06612333
Title: Evaluation of the French Version of the PEERS Social Skills Training Program for Adolescents With Rare Neurodevelopmental Disorders / PEERS-MRND
Brief Title: Evaluation of the French Version of the PEERS Social Skills Training Program for Adolescents With Rare Neurodevelopmental Disorders
Acronym: PEERS-MRND
Status: Completed | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HJ-23-PEERS-MRND
Record Dates: First submitted 2024-04-26; First posted 2024-09-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Neurodevelopmental Disorders; Rare Diseases
MeSH Terms: conditions — Neurodevelopmental Disorders; Rare Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Inclusion criteria:
  * Aged between 12 and 30 years, included at the start of the social skills program.
  * Patients with rare neurodevelopmental diseases
  * Patients benefiting from the social skills program
  * Appropriate level of verbal elaboration
  * Patient with a family member or a friend also participating in the social skills program
  Non-inclusion criteria :
  * Opposition of the patient or, if a minor, of his/her parents to participation in the study
  * Patient not psychiatrically stabilized: acute symptoms of anxiety, depression, psychotic disorders.
  * Severe intellectual disability
- Family member or friend: Inclusion criteria:
  * be over 18 years
  * be a close relative or friend of a patient and share in his or her daily life
  * have taken or are taking the social skills program
  Non-inclusion criteria :
  - Opposition to participation in the study

SUMMARY:
Adolescents and young adults with rare neurodevelopmental disorders are at risk of developing psychiatric pathologies during the transition to adulthood. Loneliness and lack of social relationships can lead to anxiety and depression in adolescents and young adults with rare neurodevelopmental disorders. Anxiety and depression are major risk factors for the transition to psychiatric symptoms in adulthood. The improvement of social skills and the positive evolution of social relationships in adolescents and young adults with rare neurodevelopmental disorders can lead to a reduction in the risk factors for anxiety and depression. It therefore seems essential to evaluate the evolution of social skills in this population of young adults under the care of the social skills program, PEERS, in France to assess the overall benefit of the program, particularly in this population of young people with rare neurodevelopmental disorders.

ELIGIBILITY:
Inclusion criteria:

* Aged between 12 and 30 years, included at the start of the social skills program.
* Patients with rare neurodevelopmental diseases
* Patients benefiting from the social skills program
* Appropriate level of verbal elaboration
* Patient with a family member or a friend also participating in the social skills program

Non-inclusion criteria :

* Opposition of the patient or, if a minor, of his/her parents to participation in the study
* Patient not psychiatrically stabilized: acute symptoms of anxiety, depression, psychotic disorders.
* Severe intellectual disability

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will focus on data from 40 patients with rare neurodevelopmental disorders and their 40 relatives/friends.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Assessment of social skills in adolescents and young adults with rare neurodevelopmental diseases participating in the social skills program | 2023 - 2025
  Quality of Play Questionnaire-Adolescent (QPQ-A) (QSQP in French)
Assessment of social skills in adolescents and young adults with rare neurodevelopmental diseases | 2023 - 2025
  Friendship Quality Scale (FQS)
Assessment of social skills in adolescents and young adults with rare neurodevelopmental diseases | 2023 - 2025
  Social Anxiety Scale for Adolescent (SAS-A)
Assessment of social skills in adolescents and young adults with rare neurodevelopmental diseases | 2023 - 2025
  Loneliness and Social Dissatisfaction Scale (L&SD)
Assessment of social skills in adolescents and young adults with rare neurodevelopmental diseases | 2023 - 2025
  Test of Adolescent Social Skills Knowledge (TASSK)
Assessment of social skills in adolescents and young adults with rare neurodevelopmental diseases | 2023 - 2025
  Self-Assessment of Conversational Skills (AHC)
Assessment of social skills in adolescents and young adults with rare neurodevelopmental diseases | 2023 - 2025
  Beck Youth Inventories (BYI)

CONTACTS AND LOCATIONS:
Locations (1):
- Necker - Enfants Malades Hospital, Paris, Île-de-France Region, France